CLINICAL TRIAL: NCT01467596
Title: Effects of Age on Minimum Effective Volume of Local Anesthetic for Ultrasound-guided Supraclavicular Brachial Plexus Block (US-SCB)
Brief Title: Ultrasound-guided Supraclavicular Brachial Plexus Block in Elderly
Acronym: US-SCB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Šarić, Jadranka Pavičić, M.D. (Individual)
Responsible Party: Principal Investigator, Jadranka Pavičić Šarić, Effects of Age on Minimum Effective Volume of Local Anesthetic for Ultrasound-guided Supraclavicular Brachial Plexus Block (US-SCB), Šarić, Jadranka Pavičić, M.D.
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT 2011-005432-26
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Arm Injuries; Anesthesia
Keywords: Ultrasound; Brachial block; Levobupivacaine; Minimum; Volume; Minimum volume of Levobupivacaine 0,5%
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly population (Experimental): MEAV50, MEAV95 Onset and duration of sensory and motor blockade
  Interventions: Device: Elderly population, Middle aged population
- Middle aged population (Active Comparator): MEAV50, MEAV95 Onset and duration of sensory and motor blockade
  Interventions: Device: Elderly population, Middle aged population

INTERVENTIONS:
Device: Elderly population, Middle aged population — The study method is a step-up/step-down sequence model where the dose of local anesthetic for the following patient is determined by the outcome of the preceding block. The starting dose of 50:50 mixture of 0.5% levobupivacaine and 2% lidocaine is 30 mL. In the case of block failure, the dose will be increased by 5 mL. Conversely, block success will result in a reduction in dose by 5 mL. A blinded assistant will assess sensory and motor blockade in each nerve territory ( the median, radial, ulnar and musculocutaneous) at 5-min intervals up to 30 min after completion of US-SCB. Effective US-SCB will be defined as complete sensory blockade in the distribution of the radial, ulnar, median and musculocutaneous nerve.
  Other Names: Levobupivacaine 0.5%; Lidocaine 2%

SUMMARY:
The aim of this study is to determine the minimum effective volume of local anesthetic (50:50 mixture of 0.5% levobupivacaine and 2% lidocaine) required to produce an effective US-SCB for surgical anesthesia in 50% of patients and to calculate the effective volume required to produce an effective US-SCB in 95% of the patients (MEAV95) in elderly group (>65 years) and in middle aged group (<45years) of patients.

DETAILED DESCRIPTION:
We believe that known data regarding the minimum anesthetic volume required for effective US-SCB from middle age population can not be applicable to the elderly population since our preliminary data, presented at Euroanesthesia meeting in Amsterdam, 2011, and published in abstract form in the European Journal of Anaesthesiology, showed that involutional changes of brachial plexus in elderly, assessed by measuring the cross-sectional area (CSA) of brachial plexus at the first rib, allowed a 35% reduction in local anesthetic volume for an effective US-SCB for surgical anesthesia in elderly patients in comparison with the younger patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 - 3 elderly patients (>65 years) scheduled for hand surgery
* ASA 1-3 middle aged patients (<45 years)

Exclusion Criteria:

* Cognitive impairment
* Coagulopathy
* Allergy to local anesthetics
* Infection at the puncture site,
* Body mass index > 35 kg/m2

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Ultrasound-guided Supraclavicular Brachial Plexus Block in Elderly | A blinded Assistant assess sensory and motor blockade in a 5-min intervals up to 30 minutes
  Determining the minimum effective volume of a 50:50 mixture of levobupivacaine 0.5% and lidocaine 2% for successful supraclavicular brachial plexus block for hand surgery in 50% of elderly patients (MEAV50) and to calculate the effective volume in 95% of the elderly patients (MEAV95) as compared with control group (middle aged patients).

SECONDARY OUTCOMES:
Ultrasound-guided Supraclavicular Brachial Plexus Block in... | A blinded Assistant assess onset (in a 5-min intervals up to 30 minutes after completion of US-SCB) ) and duration of sensory and motor blockade (in a 30-min intervals after the completion of surgery).
  Sensory and motor block onset time and duration for each nerve (median, radial, ulnar and musculocutaneous) and for the group.

CONTACTS AND LOCATIONS:
Overall Officials: Jadranka Pavičić Šarić, MD, Principal Investigator
Locations (2):
- Croatia (2):
  - University Hospital Merkur, Zagreb, City of Zagreb
  - University Hospital Merkur, Zagreb, Croatia

REFERENCES:
- [Result] Tomulic K, Pavicic Saric J, Acan I.Effect of age on anaesthetic volume for ultrasound guided supraclavicular brachial plexus block: 8AP2-8 June 2011 - Volume 28 - Issue - p 113 European Journal of Anaesthesiology